CLINICAL TRIAL: NCT05246215
Title: Diagnostic Values of Galectin-3, Soluble ST2 and BNP in Predicting the Clinical Outcome of ST-Segment Elevation Myocardial Infarction Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Khalifa Mohamed Abdelzaher, Resident doctor., Assiut University
Other Study IDs: DV_Gal_3,sST2
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: ST Elevation Myocardial Infarction; HF - Heart Failure; Stable Angina
Keywords: Galectin-3
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Heart Failure; Angina, Stable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- STEMI group.: 60 participants of patients with STEMI treated with primary percutaneous coronary intervention (pPCI).
- healthy group.: 15 participants of healthy people as a case control.
- Stable angina group.: 15 participants of patients stable angina

SUMMARY:
An acute ST-elevation myocardial infarction occurs due to occlusion of one or more coronary arteries, causing transmural myocardial ischemia which in turn results in myocardial injury or necrosis. Acute myocardial infarction (AMI) may lead to the development of heart failure (HF). Accessible diagnostic tools commonly used in HF such as natriuretic peptides and (NYHA) classiﬁcation reﬂect already overt clinical HF. Troponin and creatine kinase reﬂect myocardial damage, but their usefulness in predicting long-term LVR is limited. Recent guidelines on HF management stressed that HF onset may be delayed or prevented through certain Interventions, such as pharmacotherapy ,post infarction rehabilitation, or modiﬁcation of HF risk factors. Therefore, it is important to identify potential markers, which would be more informative of HF preclinical stages to recognize patients with an increased risk of HF onset, and to start treatment in advance (1) Gal-3 participates in inﬂammation and pro ﬁbrotic pathways, while sST2 is a biomarker of inﬂammation, cardiac mechanical strain, and tissue ﬁbrosis, both of which may predict LVR (2).

sST is a biomarker of inﬂammation, cardiac mechanical strain, and tissue ﬁbrosis(3).

B_type natriuretic peptide (BNP) is elevated in acute myocardial infarction and is a quantitative biochemical marker related to the extent of infarction and left ventricular systolic dysfunction(4).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Hospital admission due to ﬁrst-time STEMI treated with pPCI.

Exclusion Criteria:

* History of previous acute coronary syndrome, Previously diagnosed HF or asymptomatic LV dysfunction with LVEF <50% or previously diagnosed signiﬁcant valvular disease or any other previously diagnosed structural heart disease Severe renal dysfunction, Severe liver disease, Chronic inﬂammatory disease, Current neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Assuit University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
investigate the association of Gal-3, sST2 and BNP concentrations and the development of clinically overt HF in patients after ST-segment elevation myocardial infarction (STEMI) treated with primary percutaneous coronary intervention | 7 months